CLINICAL TRIAL: NCT00494741
Title: A Randomized, Prospective, Multicenter Trial to Compare the Effect on Chronic Allograft Nephropathy Prevention of Mycophenolate Mofetil Versus Azathioprine as the Sole Immunosuppressive Therapy for Kidney Transplant Recipients
Brief Title: MMF vs. AZA for Kidney Transplantation
Acronym: ATHENA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATHENA; 2006-005604-14 (EudraCT Number)
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mycophenolate mofetil (Experimental)
  Interventions: Drug: mycophenolate mofetil
- azathioprine (Experimental)
  Interventions: Drug: azathioprine

INTERVENTIONS:
Drug: mycophenolate mofetil — Patients randomized in this group will receive 750 mg of MMF per os twice a day starting on the day of transplant. MMF dose will be reduced in case of white blood cell count lower than 2,000/mm3 and whenever deemed clinically appropriate.
  Arms: mycophenolate mofetil
Drug: azathioprine — Patients randomized in this group will receive 75 mg of AZA per os (or 125 mg if body weight > 75 kg) once a day starting on the day of transplant. AZA dose will be reduced in case of white blood cell count lower than 2,000/mm3 and whenever deemed clinically appropriate.
  Arms: azathioprine

SUMMARY:
The Mycophenolate Steroid Sparing (MYSS) study demonstrated that, in the setting of a maintenance immunosuppressive regimen without steroids, mycophenolate mofetil (MMF) and azathioprine (AZA) provided the same efficacy in preventing acute rejection episodes and allograft dysfunction in kidney transplant recipients. Induction therapy with basiliximab combined with low-dose thymoglobulin (RATG), through a transient depletion/inhibition of T lymphocytes, allows further reducing the need for maintenance immunosuppression.

Aim of the present study is to assess whether under this induction strategy MMF and AZA are equally effective in preventing acute rejection and chronic allograft nephropathy (CAN), even after cyclosporine (CsA) withdrawal.

Two-hundred-twenty-four kidney transplant recipients from deceased donors given induction therapy with two 20 mg basiliximab injections 4 days apart and a seven-day course of RATG (0.5 mg/kg/day), will be randomly allocated on a 1:1 basis to 3-year treatment with low-dose MMF or AZA, added-on CsA maintenance therapy. At 1 year, rejection-free patients with no evidence of tubulitis at kidney biopsy will withdraw CsA and will have a kidney biopsy 3 year post-transplant for evaluating the presence and severity of CAN. Should the cumulative incidence of acute rejection exceed 15% during CsA withdrawal the study will be stopped. Should the incidence differ by >30% between the two treatment arms, all patients will be given the most effective treatment and the follow up will be continued. A final biopsy will be repeated 4 years post-transplant.

Most patients are expected to be effectively maintained on single drug immunosuppression, which implies less steroid- and CsA- related complications and treatment costs. MMF is expected to prevent CAN more effectively than AZA. However, should AZA be more or as effective compared to MMF, at study end all patients could be shifted to AZA, that is 15-fold less expensive than MMF. Extended to clinical practice, these findings should translate in improved patient care and major cost-savings for the Health Care System.

DETAILED DESCRIPTION:
INTRODUCTION The introduction of triple-therapy regimens that include a calcineurin inhibitor, steroids, and azathioprine (AZA) or mycophenolate mofetil (MMF) greatly reduced the risk of acute rejection in renal transplantation. However, the long-term use of both calcineurin inhibitors and steroids is associated with serious toxicities that ultimately impact patient and graft survival. Minimisation of chronic immunosuppression is therefore of paramount importance to improve patient and graft survival. Thus, the quest for strategies inducing specific immune hyporesponsiveness or even tolerance - ideally via short-term interventions that would target only the pathogenic immune response and leave the protective host immune response unimpaired - has provided a "holy grail" for transplant immunologists.

We recently found that induction therapy with basiliximab and lower (about one fourth) than conventional doses of Rabbit Anti-human Thymocyte Globulin (RATG), combined to low-dose CsA and MMF maintenance therapy, allowed ineffective prevention of acute rejection without steroids. Of note, unlike induction protocols with "standard" RATG doses, the above regimen was extremely well tolerated, avoided the risk of acute cytolysis reactions, reduced the incidence of immuno-hemolytic anemia and the need for red blood cell transfusions. Moreover, this approach did not increase the risk of CMV reactivations or lymphoproliferative disorders, even as compared to standard triple immunosuppressive regimens without induction therapy.

The doses of CsA employed in the above protocol were about half the doses currently used in clinical practice. However, even these very low doses have been reported to have a significant toxicity that, in the long-term, may adversely affect the graft function and survival. Thus, implementing innovative immunosuppressive strategies allowing to early and safely withdraw calcineurin inhibitor therapy might have major clinical implications in term of improved kidney function and long term survival. This would also avoid the adverse effects of chronic CsA therapy on arterial blood pressure, lipid profile and blood glucose that, altogether, remarkably increase the overall cardiovascular risk in these patients.

To this purpose, induction therapy with basiliximab plus low-dose RATG might help inducing a condition of reduced immuno-responsiveness that might allow to sequentially withdraw steroids and CsA without adversely affect the outcome of the graft.

Evidence that MMF suppresses the production of anti-HLA antibodies, inhibits the recruitment of mononuclear cells into the allograft, as well as the proliferation of arterial smooth muscle cells, has been taken to suggest that MMF might play an important protective effect against the development and progression of CAN. Thus, an immunosuppressive regimen based on low-dose MMF as sole antirejection drug not only would avoid chronic toxicity of steroids, and calcineurin inhibitors, but would also limit the risk of CAN, the main cause of allograft loss in the long-term. On the other hand, however, the Mycophenolate Steroid Sparing (MYSS) trial found that AZA was as effective as MMF in preventing acute allograft rejection in CsA-treated kidney transplant recipients, even after steroid withdrawal. Since acute allograft rejection is one of the strongest predictor of CAN, these findings can be taken to suggest that, in the long-term, AZA might share with MMF also a similar protective effect against the development of CAN. Moreover, it must be emphasized that chronic CsA nephrotoxicity is a major component of CAN. Thus, the prevalence and severity of CAN may be reduced in patients on CsA-free immunosuppressive regimens. In this clinical setting, the benefits of MMF against the development of CAN might not appreciably exceed those of AZA. Should this be the case, AZA might confer the same benefits of MMF, but at remarkably lower costs since, at equivalent doses, AZA is about 15 times less expensive than MMF.

Regardless of the above, MMF or AZA monotherapy would avoid or limit most of the complications of chronic immunosuppressive regimens including steroids and calcineurin inhibitors, such as metabolic, osteomuscular and cardiovascular diseases, cancer and opportunistic infections.

AIMS Primary To compare the incidence of CAN 3 years post-transplantation in patients receiving induction therapy with basiliximab and low-dose RATG and randomized to maintenance immunosuppression with low-dose MMF or AZA monotherapy.

Secondary

1. year

   * To assess the overall cumulative incidence (regardless of randomization) of acute rejections and of tubulitis at 1-year histology evaluation
   * To compare the cumulative incidence of acute rejections and of tubulitis in the two treatment groups
2. years

   * To assess the overall cumulative incidence (regardless of randomization) of biopsy-proven acute rejections during CsA tapering
   * To compare the cumulative incidence of biopsy-proven acute rejections in the two treatment groups
3. years

   * To assess the overall incidence (regardless of treatment randomization) of CAN and the possible relationships between the histology changes at 3 years and the histology findings at pre-transplant (baseline) kidney evaluation or previous acute rejection episodes observed before or after CsA withdrawal
   * To asses the global (vascular, glomerular and tubular-interstitial) score of chronic histology changes compared to baseline in the study group as a whole, in the two treatment arms and within the two subgroups completing or not completing CsA withdrawal
4. years

   * To assess patient and graft survival and function, incidence of CAN, and possible relationships between the histology changes at 4 years and the histology findings at baseline and at 3 years post-transplant, or previous acute rejection episodes observed before or after CsA withdrawal
   * To compare overall patient and graft survival and function, incidence of CAN and the global histology score in the two treatment groups.

DESIGN Two-hundred-twenty-four kidney transplant recipients from deceased donors given induction therapy with two 20 mg basiliximab injections 4 days apart, a seven-day course of RATG (0.5 mg/kg/day) and intravenous methylprednisolone for six days, will be randomly allocated on a 1:1 basis to 3-year treatment with low-dose MMF or AZA, added-on CsA maintenance therapy. At 1 year, rejection-free patients with no evidence of tubulitis at kidney biopsy will progressively taper/withdraw CsA and will have a kidney biopsy 3 year post-transplant for evaluating the presence and severity of CAN. Should the cumulative incidence of acute rejection exceed 15% during CsA withdrawal the study will be stopped. Should the incidence differ by >30% between the two treatment arms, all patients will be given the most effective treatment and the follow up will be continued. A final biopsy will be repeated 4 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years or more;
* First single or double kidney transplant from deceased donors;
* Written informed consent.

Exclusion Criteria:

* Specific contraindications to RATG therapy such as severe leucopenia (WBC<2000/mm3);
* High immunological risk - such as second transplant recipients or those who have a panel reactivity > 10%;
* History of malignancy (except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully;
* Evidence of active hepatitis C virus, hepatitis B virus or human acquired immunodeficiency virus infection;
* Any chronic clinical conditions that may affect completion of the trial or confound data interpretation;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial;
* Evidence of an uncooperative attitude;
* Any evidence that patient will not be able to complete the trial follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2007-05; Primary Completion 2016-07 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of biopsy-proven CAN at 3 years follow-up in patients completing CsA withdrawal in the two treatment groups (end phase B). | At 3 years follow-up.

SECONDARY OUTCOMES:
- To assess the overall incidence of acute rejections at 1 and 2 years. - To assess the overall incidence of CAN at 3 years. - To assess graft and patient survival at 4 years. | At 1,2,3 and 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (6):
- Italy (6):
  - Hospital "Azienda Ospedaliera Ospedali Riuniti di Bergamo" Unit of Neprology and Dialysis, Bergamo
  - Hospital "Spedali Civili" - Unit of Nephrology and Dialysis, Brescia
  - Hospital "Niguarda Cà Granda", Milan
  - Hospital "Azienda Ospedaliera di Padova" -, Padua
  - Policlinico Gemelli, Roma
  - Hospital "Az. Ospedaliero-Univeristaria S. Maria della Misericordia, Udine

REFERENCES:
- [Derived] Ruggenenti P, Cravedi P, Gotti E, Plati A, Marasa M, Sandrini S, Bossini N, Citterio F, Minetti E, Montanaro D, Sabadini E, Tardanico R, Martinetti D, Gaspari F, Villa A, Perna A, Peraro F, Remuzzi G. Mycophenolate mofetil versus azathioprine in kidney transplant recipients on steroid-free, low-dose cyclosporine immunosuppression (ATHENA): A pragmatic randomized trial. PLoS Med. 2021 Jun 24;18(6):e1003668. doi: 10.1371/journal.pmed.1003668. eCollection 2021 Jun. PMID 34166370
- [Derived] Cravedi P, Mannon RB, Remuzzi G. Lymphocyte depletion for kidney transplantation: back to the past? Nat Clin Pract Nephrol. 2008 Oct;4(10):534-5. doi: 10.1038/ncpneph0914. Epub 2008 Aug 26. No abstract available. PMID 18725917